CLINICAL TRIAL: NCT02415127
Title: Randomized, Multicenter, Double-Blind, Placebo-Controlled, Efficacy, Safety, and Pharmacokinetic Study of ACTIMMUNE® (Interferon γ-1b) in Children and Young Adults With Friedreich's Ataxia
Brief Title: Safety, Tolerability and Efficacy of ACTIMMUNE® Dose Escalation in Friedreich's Ataxia
Acronym: STEADFAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZNP-ACT-301
Record Dates: First submitted 2015-02-12; First posted 2015-04-14 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Friedreich's Ataxia
Keywords: Interferon gamma
MeSH Terms: conditions — Friedreich Ataxia | interventions — interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Interferon γ-1b (Experimental): Approximately 45 participants will receive subcutaneous (SC) doses of ACTIMMUNE® 3 times a week (TIW) for a total of 26 weeks.
  Interventions: Drug: Interferon γ-1b
- Placebo (Placebo Comparator): Approximately 45 participants will receive SC doses of placebo TIW for a total of 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon γ-1b — The study drug dose is planned to be escalated on a weekly basis over the first 4 weeks of treatment (from 10 µg/m² to 25, 50, and 100 µg/m²). The dose may be reduced, interrupted, or held based on tolerability. By Week 13, all participants are to be on a stable tolerated dose of study drug in order to continue study participation; the dose may not be further increased after week 13, however, it may be reduced on a case-by-case basis to manage drug-related adverse events (AEs).
  Other Names: ACTIMMUNE®
  Arms: Interferon γ-1b
Drug: Placebo — The volume of placebo is planned to correspond with volume of study drug that would be given to the participant if the participant was randomized to the study drug arm.
  Arms: Placebo

SUMMARY:
The purpose of this phase 3 randomized, multi-center, double-blind, placebo-controlled study is to evaluate the efficacy and safety of ACTIMMUNE® (interferon-γ 1b) in the treatment of Friedreich's Ataxia (FA) and to evaluate the pharmacokinetic (PK) characteristics of ACTIMMUNE® in FA patients.

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and child assent, if applicable.
* FA confirmed by genetic testing with two expanded guanine-adenine-adenine (GAA) repeats.
* FA functional stage of >1 to <5 and ability to walk 25 feet with or without an assistive device.
* Male or female subject between the ages of 10 and 25 years, inclusive.
* If female, the subject is not pregnant or lactating or intending to become pregnant during the study, or within 30 days after the last dose of study drug. Female subjects of child-bearing potential must have a negative serum pregnancy test result at Screening, a negative urine pregnancy test result at Baseline, and agree to use a reliable method of contraception throughout the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* Any unstable illness that in the investigator's opinion precludes participation in the study.
* Use of any investigational product within 30 days prior to randomization.
* A history of substance abuse.
* Presence of clinically significant cardiac disease (as determined by the investigator based on electrocardiogram [ECG] and echocardiogram results at Screening). Specifically, an ejection fraction of <40% or a prolonged QT interval (>50% of cycle duration) will result in exclusion. If the investigator notes any other clinically significant abnormalities on the ECG or echocardiogram, the subject may be eligible if they are provided clearance from a cardiologist.
* History of hypersensitivity to interferon (IFN)-ɣ or E. coli-derived products.
* Presence of moderate or severe renal disease (estimated creatinine clearance <50 mL/min) or hepatic disease (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2x the upper limit of normal) as evidenced by laboratory results at Screening.
* Clinically significant abnormal white blood cell count, hemoglobin, or platelet count as evidenced by laboratory test results at Screening.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - University of California, Los Angeles Neurology Clinic, Los Angeles, California
  - University of Florida - Clinical Research Center, Gainesville, Florida
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon γ-1b: Subcutaneous (SC) doses of ACTIMMUNE® 3 times a week (TIW) for a total of 26 weeks.
- Placebo: SC doses of placebo TIW for a total of 26 weeks.
Period: Overall Study
Arm/Group | Interferon γ-1b | Placebo
Started | 47 | 45
Completed | 46 | 45
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interferon γ-1b: SC doses of ACTIMMUNE® TIW for a total of 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Interferon γ-1b | Placebo | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (4.41) | 16.1 (3.75) | 16.3 (4.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in the Friedreich's Ataxia Rating Scale (FARS)-mNeuro Score
Description: The FARS assessment includes neurological signs that specifically reflect neural substrates affected in FA. Based on a neurological examination, bulbar, upper limb, lower limb, peripheral nerve, and upright stability/gait functions were assessed. The FARS-mNeuro score excludes the peripheral nervous system subscale score and the facial and tongue atrophy and fasciculations from the bulbar subscale score. Scores range from 0 (normal) to 93 (most impairment). A negative change from baseline is an improvement.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat (ITT) Population: All randomized participants with a valid baseline (including Screening) and at least 1 valid post baseline measurement in the primary efficacy outcome (FARS-mNeuro) and at Week 26. A valid FARS-mNeuro score was defined as no missing values in the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon γ-1b | Placebo
Number analyzed (Participants) | 46 | 44
units on a scale | -0.6 (4.61) | -1.0 (4.41)
Statistical Analysis 1: Comparison: Interferon γ-1b vs Placebo; The primary and secondary efficacy endpoints were tested in a hierarchical manner. Each endpoint was tested in sequential order and the current endpoint must have shown statistical significance (p < 0.05) prior to performing testing the next endpoint. The primary endpoint, FARS-mNeuro, was to be tested first, followed by the key secondary endpoint, ADL, followed by the other secondary endpoints, T25FW, FARS-mNeuro responder rate, and FARStot; Test type: Superiority; p = 0.5442, ANCOVA — From a repeated-measures ANCOVA with fixed effects of treatment, visit, and treatment*visit with baseline score and investigative site as covariates using an unstructured covariance matrix, testing ACTIMMUNE® vs placebo

2. Secondary Outcome: Change From Baseline to Week 26 in Activities of Daily Living (ADL) Score
Description: Participants and/or their caregivers rated 9 areas of daily living skills (speech, swallowing, cutting food and handling utensils, dressing, personal hygiene, falling, walking, quality of sitting position, and bladder function) on a 5-point scale (0=normal, 4=greatest loss of function) with allowable increments of 0.5 if the participant or caregiver strongly felt that a task falls between 2 scores. ADL scores can range from 0 (normal) to 36 (greatest loss of function). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population: All randomized participants with a valid baseline (including Screening) and at least 1 valid post baseline measurement in the primary efficacy outcome (FARS-mNeuro) and ADL data at Baseline and Week 26. A valid FARS-mNeuro score was defined as no missing values in the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon γ-1b | Placebo
Number analyzed (Participants) | 46 | 45
units on a scale | 0.64 (2.938) | 0.01 (2.595)

3. Secondary Outcome: Change From Baseline at Week 26 in Timed 25-Foot Walk (T25FW)
Description: The T25FW is a quantitative measure of lower extremity function. Participants are directed to 1 end of a clearly marked 25-foot course and instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the participant walk back the same distance, and the score for the test is the average of the 2 walks (after reciprocal transformation). Participants may use assistive devices when performing this task, with the same assistive device used at each assessment. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population: All randomized participants with a valid baseline (including Screening) and at least 1 valid post baseline measurement in the primary efficacy outcome (FARS-mNeuro), and T25FW data at Baseline and Week 26. A valid FARS-mNeuro score was defined as no missing values in the questionnaire.
Measure: Mean (Standard Deviation); unit: 1/seconds
Arm/Group | Interferon γ-1b | Placebo
Number analyzed (Participants) | 44 | 42
1/seconds | -0.006 (0.0247) | -0.003 (0.0181)

4. Secondary Outcome: Number of FARS-mNeuro Responders and Non-Responders at Week 26
Description: A participant was considered a responder if they had an improvement (decrease) of at least 3 points from Baseline at Week 26 for the FARS-mNeuro score. The FARS assessment includes neurological signs that specifically reflect neural substrates affected in FA. Based on a neurological examination, bulbar, upper limb, lower limb, peripheral nerve, and upright stability/gait functions were assessed. The FARS-mNeuro score excludes the peripheral nervous system subscale score and the facial and tongue atrophy and fasciculations from the bulbar subscale score. Scores range from 0 (normal) to 93 (most impairment).
Time Frame: Week 26
Population: ITT Population: All randomized participants with a valid baseline (including Screening) and at least 1 valid post baseline measurement in the primary efficacy outcome (FARS-mNeuro) and data at Week 26. A valid FARS-mNeuro score was defined as no missing values in the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Interferon γ-1b | Placebo
Number analyzed (Participants) | 46 | 44
Participants
  Responder | 14 | 16
  Non-responder | 32 | 28

5. Secondary Outcome: Change From Baseline to Week 26 in Total Friedreich Ataxia Rating Scale Score (FARStot)
Description: The FARS assessment includes neurological signs that specifically reflect neural substrates affected in FA. Based on a neurological examination, bulbar, upper limb, lower limb, peripheral nerve, and upright stability/gait functions are assessed. FARStot scores range from 0 (normal) to 125 (most impairment). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 26
Population: ITT Population: All randomized participants with a valid baseline (including Screening) and at least 1 valid post baseline measurement in the primary efficacy outcome (FARS-mNeuro) and FARStot data at Baseline and Week 26. A valid FARS-mNeuro score was defined as no missing values in the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon γ-1b | Placebo
Number analyzed (Participants) | 46 | 44
units on a scale | -0.2 (5.53) | -0.6 (5.19)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are presented. Adverse events (AEs) occurring or worsening after the dose on Day 1 through the end of the study (Week 26) were considered TEAEs. Serious TEAEs were collected through 2 weeks after study discontinuation (Week 28).
Arm/Group | Interferon γ-1b | Placebo
Serious Adverse Events (participants affected / at risk) | 1/47 | 2/45
Other Adverse Events (participants affected / at risk) | 45/47 | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon γ-1b (N=47) | Placebo (N=45)
Chest pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon γ-1b (N=47) | Placebo (N=45)
Neutropenia (Blood and lymphatic system disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 18 | 11
Vomiting (Gastrointestinal disorders) | 3 | 4
Chills (General disorders) | 6 | 2
Fatigue (General disorders) | 4 | 8
Injection site bruising (General disorders) | 5 | 5
Injection site erythema (General disorders) | 7 | 1
Injection site pain (General disorders) | 5 | 3
Injection site pruritus (General disorders) | 4 | 1
Pain (General disorders) | 4 | 2
Pyrexia (General disorders) | 7 | 8
Nasopharyngitis (Infections and infestations) | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 5 | 4
Excoriation (Injury, poisoning and procedural complications) | 3 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 3
Joint injury (Injury, poisoning and procedural complications) | 3 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 4
Neutrophil count decreased (Investigations) | 4 | 0
White blood cell count decreased (Investigations) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 6 | 4
Headache (Nervous system disorders) | 24 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .